CLINICAL TRIAL: NCT01472406
Title: Artificial Pancreas Device Feasibility Study for Type 1 Diabetes Patients Using Model-predictive Control and Health Monitoring System Algorithms With an Approved Subcutaneous Insulin Delivery Pump and Subcutaneous Continuous Glucose Monitor
Brief Title: Feasibility Study Using Zone-MPC Controller (Zone-Model Predictive Control) and Health Monitoring System (HMS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: University of California, Santa Barbara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DK085628
Record Dates: First submitted 2011-10-27; First posted 2011-11-16 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; closed-loop artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed-loop session (Experimental): The study consists of an evaluation of the Sansum Closed-loop Artificial Pancreas Device, insulin infusion pump, Continuous Glucose Monitor, zone-Model Predictive Control algorithm, and a Safety Health Monitoring System. during a 24-hour closed-loop in a clinic environment (Sansum Diabetes Research Institute, Santa Barbara, CA).
  Interventions: Device: Sansum Closed-Loop Artificial Pancreas; Device: Insulin infusion pump; Device: Continuous Glucose Monitor; Device: zone-Model Predictive Control algorithm; Device: Safety Health Monitoring System

INTERVENTIONS:
Device: Sansum Closed-Loop Artificial Pancreas — The Sansum Closed-loop Artificial Pancreas Device is the infrastructure that allows communication between the insulin pump, the CGM, the zone-MPC, and the HMS.
  Other Names: Sansum AP
Device: Insulin infusion pump — The insulin pump, which has received 510k clearance (K080639), delivers insulin subcutaneously through an infusion set.
Device: Continuous Glucose Monitor — The CGM, which is an approved device (P050012), measures interstitial glucose.
  Other Names: CGM
Device: zone-Model Predictive Control algorithm — The zone-MPC predicts future glucose values, based on CGM data, to regulate blood glucose level by increasing, decreasing, or stopping insulin infusion via an insulin infusion pump.
  Other Names: zone-MPC
Device: Safety Health Monitoring System — The HMS predicts future glucose values, based on CGM data, to warn the Sansum Closed-loop Artificial Pancreas Device of values below 70 mg/dL.
  Other Names: HMS

SUMMARY:
This clinical trial is a feasibility study to assess the performance of an Artificial Pancreas (AP) device using the Artificial Pancreas System (APS©) platform for subjects with type 1 diabetes. The device is a closed-loop between a DexCom™ SEVEN® PLUS (DexCom™ Corp, San Diego, CA) continuous glucose monitor (CGM) and a OneTouch® Ping® Glucose Monitoring System (Animas Corp, Westchester, PA) subcutaneous insulin delivery pump (CSII). The AP device is controlled by a zone-Model Predictive Control (zone-MPC) algorithm augmented by a safety algorithm named the Health Monitoring System (HMS). The clinical study will include 12 to 20 adults subjects aged 21 to 65 years old.

DETAILED DESCRIPTION:
The study consists of an evaluation of the Artificial Pancreas device during a 24-hour closed-loop in a clinic environment (Sansum Diabetes Research Institute, Santa Barbara, CA). The 24-hour period includes:

* 2 unannounced meals (evening dinner and breakfast);
* 1 period of 30 minutes of exercise at 50% of the predicted heart rate reserve (HRR) preceded with a snack and followed by a snack 3 hours later (on Day 2);
* complete night from 12:00 am to 7:00 am; The subject will arrive at approximately 4:00 pm to the CRC (clinical research center), the closed-loop will be initiated at approximately 4:30 pm that same day and continued until 4:30 pm the next day. A physician will be monitoring the patient with the artificial Pancreas (AP) device at all time.

The proposed study will evaluate the performance of the AP device in predicting the fall and rise of glucose values and in regulating insulin delivery to mitigate extreme blood glucose variations during the following challenges:

* following unannounced meals,
* during a nocturnal period, and
* during a period of active exercise.

The goal is to demonstrate that the AP device is able to maintain the subject blood glucose within a safe range at all times. One of the objectives of the study will be to measure the percent of time spent in the following zones:

* [80-140] mg/dL at all times unless described otherwise
* [80-140] mg/dL during the nocturnal period
* [70-180] mg/dL postprandial, for 5 hours following the unannounced meals
* [70-150] mg/dL during and for 3 hours following exercise It is anticipated that following the planned challenges, glucose value might increase temporarily beyond those ranges. These excursions will be reviewed and analyzed (value and duration) and the study will determine how the AP device mitigates those excursions and maintains glucose levels within a safe and acceptable range. The clinical study will also review any event that occur during the course of the 24-hour closed-loop: hypoglycemic events, hyperglycemic events, outside intervention, other Adverse Event, Serious Adverse Events, Unanticipated Adverse Device Effect, and device complaints for the commercial devices used. The safety of the patient will remain the primary goal. The goal of the AP device is to operate without outside intervention even when challenged by meals or exercise unless the outside intervention is requested by the Health Monitoring System (HMS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 6 months with commercially available rapid actin insulin
* The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 21 to 65 years
* For females, not currently known to be pregnant or nursing
* HbA1c between 5.0% and 10%, as measured with DCA2000 or equivalent device
* Willing to perform the calibration of the study CGMs using a finger stick only and willing to follow instructions for insulin pump and CGM wear.
* Willing to use the study CGM and study insulin pump during closed-loop.
* Able to and agrees to avoid the following medication starting 24 hours before sensor wear through completion of CRC visit: acetaminophen, prednisone, and pseudoephedrine.
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Pregnancy (as determined by a positive blood pregnancy test performed in females of childbearing capacity during screening visit and urine test at time of admission for in-patient visit) or nursing mother.
* Diabetic ketoacidosis in the past 6 months prior to enrollment requiring emergency room visit or hospitalization
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* Current treatment for a seizure disorder; Subjects with a history of seizures may be included in the study if they receive written clearance from their neurologist
* Cystic fibrosis
* Active infection
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as cognitive deficit.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation, including subjects not able to read or write.
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
* Coronary artery disease or heart failure. Subjects with a history of coronary artery disease may be included in the study if they receive written clearance from their cardiologist
* Presence of a known adrenal disorder
* Active coronary artery disease or heart failure
* Active gastroparesis
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Uncontrolled thyroid disease. Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
* Abuse of alcohol
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Current use of a beta blocker medication
* Laboratory results:

  * Hematocrit < 30% or >55%
  * A1C > 10%
  * Abnormal liver or renal function (Transaminase > 2 times the upper limit of normal, Creatinine> 1.5 mg/dL)
  * Labs drawn at screening visit or within one month prior to screening (for other purposes) will suffice for enrollment purposes related to hematocrit
* Subject has skin conditions that, in the determination of the investigator, would preclude wearing the study devices (infusion set and sensor), in the abdomen. Examples include but are not limited to: psoriasis, burns, scaring, eczema, tattoos, and significant hypertrophy at sites of device wear; any known allergy to medical adhesives.
* Current participation in another investigational trial or has previously participated to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
% of time within zone [80-140] mg/dL except 5 hours post-prandial and during exercise and 3 hours post-exercise | 24 hours
  Measures ability of AP device to maintain glucose level within a safe zone and to return to save zone following unannounced meals and exercises.

SECONDARY OUTCOMES:
% of time within zone [80-140] mg/dL during night between 12:00 am and 7:00 am | 24 hours
  Measures ability of AP device to maintain glucose level with a safe zone during the night and prevent hypoglycemia
% of time within zone [70-180] mg/dL 5 hours after unannounced evening meal, and breakfast | 24 hours
  Measures ability of AP device to react to small meal and to prevent glucose level from dangerous excursions.
% of time within zone [70-150] mg/dL during the 30 min exercise | 24 hours
  Measures ability of AP device to maintain safe glucose level during 30 minutes of non-strenuous exercise
% of time within zone [70-150] mg/dL during the 3 hours following exercise | 24 hours
  Measures ability of AP device to address exercise and to prevent glucose level from dangerous excursions

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Sansum Diabetes Research Institute; Francis J Doyle, PhD, Study Director — University of California, Santa Barbara
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

REFERENCES:
- [Derived] Harvey RA, Dassau E, Bevier WC, Seborg DE, Jovanovic L, Doyle FJ 3rd, Zisser HC. Clinical evaluation of an automated artificial pancreas using zone-model predictive control and health monitoring system. Diabetes Technol Ther. 2014 Jun;16(6):348-57. doi: 10.1089/dia.2013.0231. Epub 2014 Jan 28. PMID 24471561